CLINICAL TRIAL: NCT04691895
Title: Gastrointestinal Symptoms of SARS-CoV-2 Infection: a Prospective Multicentre Study
Brief Title: Gastrointestinal Symptoms in COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Giovanni Barbara, Professor, University of Bologna
Other Study IDs: GI-COVID19_01
Record Dates: First submitted 2020-12-09; First posted 2020-12-31 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: COVID19 Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients admitted to hospital for COVID19 disease (case group): The study cohort will be composed by consecutively enrolled COVID19 confirmed inpatients (case group)
  Inclusion criteria:
  * Signed informed consent
  * Age ≥18 years and ≤85 years
  * Consecutive COVID19 confirmed patients (COVID +ve)
  * Ability to conform to study protocol
  Exclusion criteria:
  * Patients under mechanical ventilation
  * Patients unable to report required data
  * Current diagnosis of cancer
  Interventions: Other: SARS-CoV2 infection
- Patients admitted to hospital in absence of COVID19 disease (control group): The study cohort will be composed by consecutively enrolled COVID19 negative patients hospitalized for other reasons (controls group)
  Inclusion criteria:
  * Signed informed consent
  * Age ≥18 years and ≤85 years
  * Consecutive hospitalized COVID19 negative patients (COVID -ve)
  * Ability to conform to study protocol
  Exclusion criteria:
  * Patients under mechanical ventilation
  * Patients unable to report required data
  * Current diagnosis of cancer

INTERVENTIONS:
Other: SARS-CoV2 infection — Confirmed COVID19 cases The definitions of COVID19 state are according to the WHO document released in March 2020. A person with laboratory confirmation of COVID-19 infection, irrespective of clinical signs and symptoms.
  Groups: Patients admitted to hospital for COVID19 disease (case group)

SUMMARY:
The coronavirus disease 2019 (COVID-19) initially developed at the beginning of December 2019 in Whuan, Hubei province of China has spread all over the world. Beside the most common symptoms at onset of illness including fever, fatigue, dry cough, myalgia and dyspnoea, there are less common symptoms such as headache abdominal pain, diarrhoea, nausea and vomiting. The proportion of patients complaining gastrointestinal symptoms is variable between 3,4% and 17,0%. Interestingly, the severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) RNA has been reported to be detectable in 50% of patients' stool samples and in these patients around the 50% had diarrhoea.

SARS-CoV2 transmission has been reported to be through droplets. However, mounting evidence indicates that SARS-CoV2 has a tropism for the gastrointestinal tract and is excreted with faeces. Accordingly, a faecal-oral route of transmission of the virus has been recently postulated. Indeed, SARS-CoV2 binds to host ACE 2 receptors (ACE2) to entry into cells which are abundantly expressed by intestinal epithelial cells and regulate intestinal inflammation. Taken together, this evidence could provide a rational basis for the development of gastrointestinal symptoms reported by COVID19 infected patients.

Primary aim: to evaluate the prevalence and prognosis of gastrointestinal symptoms in patients admitted to hospital for COVID19 disease Secondary aims

1. to evaluate long term consequences of COVID-19 on gastrointestinal symptoms
2. to evaluate long term consequences of COVID-19 on the development of post-infection irritable bowel syndrome (PI-IBS)
3. to evaluate long term consequences of COVID-19 on the development of post-infection dyspepsia
4. to assess the clinical and laboratory predictors (risk factors) of post-infection gastrointestinal symptom development

DETAILED DESCRIPTION:
The investigators propose a multicentre observational prospective study according to the clinical routine practice of coronavirus disease 2019 (COVID-19) patients. All patients will be clinically evaluated at admission according to standard clinical practice. All data present in the inpatient medical record will be used for the study.

The study cohort will be composed by consecutively enrolled COVID19 confirmed inpatients (case group) and COVID19 negative patients hospitalized for other reasons (controls group) referred to the participants centres from May 1, 2020.

Patient's follow up will start at discharge and will continue for 12 months.

Definitions Confirmed COVID19 cases The definitions of COVID19 state are according to the World Health Organization (WHO) document released in March 2020.

A person with laboratory confirmation of COVID-19 infection, irrespective of clinical signs and symptoms. Patients categorized as suspect or probable COVID19 cases will be excluded from enrolment.

COVID19 negative patients (controls) Consecutive COVID19 negative in-patients admitted for any clinical condition other than a primary gastrointestinal disease fulfilling the inclusion criteria.

Visits and evaluations After enrolment, all patients will be contacted telephonically at 1 month after discharge for reassessment of Gastrointestinal Symptom Rating Scale (GSRS). Subsequently, patients will be contacted every 6 months for a total of 12 months. At telephonic evaluation at 6 and 12 months after discharge patients will undergo the GSRS questionnaire, the Rome IV Diagnostic Questionnaire for Functional Gastrointestinal Disorders in Adults (R4DQ) and the hospital anxiety and depression scale (HADS) and thus the onset of PI-IBS will be recorded.

Data Management Data flow Data will be collected in custom electronic Case Report Forms (e-CRFs) on REDCap platform. System backups for data stored and records retention for the study data will be consistent with standard procedures.

Electronic Case Report Forms eCRFs are to be completed using RedCAP system. Sites will receive training and a have access to a manual for appropriate eCRF completion. eCRFs will be submitted electronically and should be handled in accordance with instructions. All eCRFs should be completed by designated, trained site staff. eCRFs should be reviewed and electronically signed and dated by the investigator or a designee.

Safety of Electronic data Data will be collected in an ad hoc electronic record storage. The creation and the management of electronic record storage will be evaluated preliminarily with institution information technology staff. Data will be collected in REDCap platform. Redcap platform is an online platform maintained in a server that is propriety of the institution. Access and data transfer from and to REDCap platform are managed under https protocol and 128-bit encryption wit SSL certificate (a secure connection with encrypted data transfer). The access at the site is allowed only for the investigators and require a user-specific password of at least 8 characters including number and special character. Redcap comes with a system of user privileges, so only the account of the principal investigator has the authorization to explore the entire dataset. The sub-investigators and data manager have limited authorizations,and can see only data that they entered personally. REDCap provider and the principal investigator guarantee that creation and management of username and password are compliant with privacy law.

The access of REDCap platform is regulated by law for protection of personal data. Administrative procedures on applications (e.g. user creation and suspension, study configuration, query creation, data mining) are pertinence of the principal investigator and his information technology support team. REDCap platform, to manage identity of people involved in the study, generates a unique identification number associated at every eCRF of the subject, that allow the investigators to maintain association with name and surname of the subject locally.

Data collected on REDCap, even if they do not allow to associate data with a specific subject or to recognize the subject, are registered in double-key SSL encryption, and maintained with AES 128 encryption. As regulated by law for protection of personal data, REDCap and the principal investigator guarantee the weekly backup of data in a password-protected storage.

Data will be accessed only by principal investigator and his support team (sub investigators), and they will have confidentiality obligation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥18 years and ≤85 years
* Consecutive COVID19 confirmed patients (COVID +ve) (case group)
* Consecutive hospitalized COVID19 negative patients (COVID -ve) (control group)
* Ability to conform to study protocol

Exclusion Criteria:

* Patients under mechanical ventilation
* Patients unable to report required data
* Current diagnosis of cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will be composed by consecutively enrolled COVID19 confirmed inpatients (case group) and COVID19 negative patients hospitalized for other reasons (controls group) referred to the participants centres from May, 1 2020. From the beginning of the study (first patient enrolled in the centre), the enrolment will last for 1 month.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of gastrointestinal symptoms in patients admitted to hospital for COVID19 disease as assessed by GSRS questionnaire | one month
  For the primary aims of the study, the presence of gastrointestinal symptoms at admission and at follow-up made 1 month after discharge will be evaluated.
  In particular, the validated Gastrointestinal Symptom Rating Scale (GSRS) questionnaire (a 7-points Likert scale) will be used to assess the prevalence of gastrointestinal symptoms.
Prognosis of gastrointestinal symptoms in patients admitted to hospital for COVID19 disease | one month
  For the prognosis, mortality rates (%) at one month will be evaluated.

SECONDARY OUTCOMES:
Long term consequences of COVID-19 on gastrointestinal symptoms on the development of post-infection (PI) irritable bowel syndrome (IBS). | 12 months
  to evaluate long term consequences of COVID-19 on the development of PI IBS, the validated Rome IV Diagnostic Questionnaire for Irritable Bowel syndrome will be used. This questionnaire translates the Rome IV diagnostic criteria into questions that can be understood and reported by patients, assisting the clinicians in arriving at a positive diagnosis. The prevalence (%) of new IBS diagnosis will be evaluated by this questionnaire.
long term consequences of COVID-19 on gastrointestinal symptoms on the development of post-infection (PI) dyspepsia. | 12 months
  to evaluate long term consequences of COVID-19 on the development of PI dyspepsia, the validated Rome IV Diagnostic Questionnaire for Dyspepsia will be used. This questionnaire translates the Rome IV diagnostic criteria into questions that can be understood and reported by patients, assisting the clinicians in arriving at a positive diagnosis. The prevalence (%) of new dyspepsia diagnosis will be evaluated by this questionnaire.
Identification of risk factors for post-infection gastrointestinal symptom development. | 12 months
  Data recorded at admission and used for the primary aims of the study will be tested as predictors of post-infection gastrointestinal symptoms onset occurring within a specific time frame using the Logistic Regression or Cox regression method. Subsequently to confirm their independent predictive value, the variables with p <0.1 will be studied in a multivariate logistic or Cox model.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barbara, MD, Principal Investigator — University of Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be collected in an ad hoc electronic record storage. The creation and the management of electronic record storage will be evaluated preliminarily with institution information technology staff. Data will be collected in REDCap platform. Data will be accessed only by principal investigator and his support team (sub investigators), and they will have confidentiality obligation.

REFERENCES:
- [Derived] Marasco G, Cremon C, Barbaro MR, Cacciari G, Falangone F, Kagramanova A, Bordin D, Drug V, Miftode E, Fusaroli P, Mohamed SY, Ricci C, Bellini M, Rahman MM, Melcarne L, Santos J, Lobo B, Bor S, Yapali S, Akyol D, Sapmaz FP, Urun YY, Eskazan T, Celebi A, Kacmaz H, Ebik B, Binicier HC, Bugdayci MS, Yagci MB, Pullukcu H, Kaya BY, Tureyen A, Hatemi I, Koc ES, Sirin G, Caliskan AR, Bengi G, Alis EE, Lukic S, Trajkovska M, Hod K, Dumitrascu D, Pietrangelo A, Corradini E, Simren M, Sjolund J, Tornkvist N, Ghoshal UC, Kolokolnikova O, Colecchia A, Serra J, Maconi G, De Giorgio R, Danese S, Portincasa P, Di Sabatino A, Maggio M, Philippou E, Lee YY, Salvi D, Venturi A, Borghi C, Zoli M, Gionchetti P, Viale P, Stanghellini V, Barbara G; GI-COVID19 study group. Post COVID-19 irritable bowel syndrome. Gut. 2022 Dec 9:gutjnl-2022-328483. doi: 10.1136/gutjnl-2022-328483. Online ahead of print. PMID 36591612
- [Derived] Marasco G, Cremon C, Barbaro MR, Salvi D, Cacciari G, Kagramanova A, Bordin D, Drug V, Miftode E, Fusaroli P, Mohamed SY, Ricci C, Bellini M, Rahman MM, Melcarne L, Santos J, Lobo B, Bor S, Yapali S, Akyol D, Sapmaz FP, Urun YY, Eskazan T, Celebi A, Kacmaz H, Ebik B, Binicier HC, Bugdayci MS, Yagci MB, Pullukcu H, Kaya BY, Tureyen A, Hatemi I, Koc ES, Sirin G, Caliskan AR, Bengi G, Alis EE, Lukic S, Trajkovska M, Hod K, Dumitrascu D, Pietrangelo A, Corradini E, Simren M, Sjolund J, Tornkvist N, Ghoshal UC, Kolokolnikova O, Colecchia A, Serra J, Maconi G, De Giorgio R, Danese S, Portincasa P, Di Stefano M, Maggio M, Philippou E, Lee YY, Venturi A, Borghi C, Zoli M, Gionchetti P, Viale P, Stanghellini V, Barbara G; and the GI-COVID19 Study Group. Prevalence of Gastrointestinal Symptoms in Severe Acute Respiratory Syndrome Coronavirus 2 Infection: Results of the Prospective Controlled Multinational GI-COVID-19 Study. Am J Gastroenterol. 2022 Jan 1;117(1):147-157. doi: 10.14309/ajg.0000000000001541. PMID 34751672